CLINICAL TRIAL: NCT02054013
Title: Prostatic Artery Embolization vs. Conventional Transurethral Prostatectomy in the Treatment of Benign Prostatic Hyperplasia: A Prospective Randomized Trial
Brief Title: Prostatic Artery Embolization vs. Conventional Transurethral Prostatectomy in the Treatment of Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Stephan Engeler (Other)
Responsible Party: Sponsor-Investigator, Daniel Stephan Engeler, Dr. med., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTU 13.030
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostatic artery embolization (Experimental): Prostatic artery embolization (PAE) has been suggested as a minimal invasive alternative procedure with rapid recovery and low morbidity
  Interventions: Procedure: Prostatic artery embolization
- Conventional monopolar transurethral prostatectomy (Other): Standard treatment
  Interventions: Procedure: monopolar transurethral prostatectomy

INTERVENTIONS:
Procedure: Prostatic artery embolization
  Arms: Prostatic artery embolization
Procedure: monopolar transurethral prostatectomy
  Arms: Conventional monopolar transurethral prostatectomy

SUMMARY:
Benign prostatic hyperplasia (BPH) is a prevalent entity, affecting over 50% of men older than 60 years. The clinical picture of the disease includes lower urinary tract symptoms such as interrupted and weak urinary stream, nocturia, urgency and leaking and even sexual dysfunction in some individuals. Medical therapy is usually the first-line treatment. However, the efficacy of drugs like alpha-blockers is limited, and as disease progresses more invasive treatment options have to be taken into consideration. In cases with moderate to severe lower urinary tract symptoms (LUTS) transurethral resection of the prostate (TUR-P) is the standard treatment. TURP, however, is limited to prostates smaller than 60-80ml and the procedure is associated with a complication rate. The cumulative short-term morbidity rate is around 11% and the necessity for surgical revision is as high as 6%. Bleeding requiring transfusions and transurethral resection syndrome represent potentially serious threats to elderly and frail patients. Prostatic artery embolization (PAE) has been suggested as a minimal invasive alternative procedure, which can be performed in an outpatient setting with rapid recovery and low morbidity.

The investigators hypothesize that PAE is non-inferior in the treatment of symptomatic BPH compared to conventional and established TUR-P.

ELIGIBILITY:
Inclusion Criteria:

* Men older than 40
* Patient must be a candidate for TURP
* Refractory to medical therapy or patient is not willing to consider (further) medical treatment
* Patient has a prostate size of at least 25 ml and not more than 80 ml, measured by ultrasound
* IPSS ≥8
* QoL ≥3
* Qmax<12 and/or urinary retention
* Written informed consent

Exclusion Criteria:

* Mild symptoms (IPSS <8)
* Severe atherosclerosis
* Severe tortuosity in the aortic bifurcation or internal iliac arteries
* Acontractile detrusor
* Neurogenic lower urinary tract dysfunction
* Urethral stenosis
* Bladder diverticulum
* Bladder stone with surgical indication
* Allergy to intravenous contrast media
* Contraindication for MRI imaging
* Preinterventionally proven adenocarcinoma of the prostate
* Renal failure (GFR<60ml/min)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
Changes in the International Prostate Symptom Score | Baseline and 12 weeks after intervention

SECONDARY OUTCOMES:
Changes of prostate volume using Magnetic Resonance Imaging | Baseline, 12 weeks and 24 months after intervention
Changes in bladder diary | Baseline and at all follow up controls
  Changes in bladder diary (difference of voids during daytime and night-time, difference voided volume, difference liquid intake, difference incontinence episodes)
Pre- and postoperative changes in C-reactive Protein, Prostate-specific antigen (PSA), serum amyloid A, Interleukin-6 and Interleukin-10 | Baseline and 1 day, 2 days, 1 and 6 weeks post intervention
Changes in urodynamic parameters | Baseline and 12 and 24 months after intervention
Duration of hospitalization post procedure | hospital discharge
Duration of post procedure catheterization | baseline and post intervention
Changes in the CPSI and IIEF | baseline and at all follow-up controls after the intervention
Procedure time and radiation parameters | after intervention
Comparison of prostate size, measured preoperatively by TRUS and MRI at baseline Comparison of prostate size, measured preoperatively by TRUS and MRI at baseline Comparison of prostate size measured by TRUS and MRI | baseline
Percentage of prostate tissue devascularized, based on contrast-enhanced MRI | 12 weeks and 24 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Engeler, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Background] Abt D, Mordasini L, Hechelhammer L, Kessler TM, Schmid HP, Engeler DS. Prostatic artery embolization versus conventional TUR-P in the treatment of benign prostatic hyperplasia: protocol for a prospective randomized non-inferiority trial. BMC Urol. 2014 Nov 25;14:94. doi: 10.1186/1471-2490-14-94. PMID 25425136
- [Background] Abt D, Hechelhammer L, Mullhaupt G, Markart S, Gusewell S, Kessler TM, Schmid HP, Engeler DS, Mordasini L. Comparison of prostatic artery embolisation (PAE) versus transurethral resection of the prostate (TURP) for benign prostatic hyperplasia: randomised, open label, non-inferiority trial. BMJ. 2018 Jun 19;361:k2338. doi: 10.1136/bmj.k2338. PMID 29921613
- [Background] Mullhaupt G, Hechelhammer L, Diener PA, Engeler DS, Gusewell S, Schmid HP, Mordasini L, Abt D. Ejaculatory disorders after prostatic artery embolization: a reassessment of two prospective clinical trials. World J Urol. 2020 Oct;38(10):2595-2599. doi: 10.1007/s00345-019-03036-7. Epub 2019 Dec 7. PMID 31813028
- [Background] Mullhaupt G, Hechelhammer L, Engeler DS, Gusewell S, Betschart P, Zumstein V, Kessler TM, Schmid HP, Mordasini L, Abt D. In-hospital cost analysis of prostatic artery embolization compared with transurethral resection of the prostate: post hoc analysis of a randomized controlled trial. BJU Int. 2019 Jun;123(6):1055-1060. doi: 10.1111/bju.14660. Epub 2019 Jan 28. PMID 30578705
- [Background] Abt D, Mullhaupt G, Hechelhammer L, Markart S, Gusewell S, Schmid HP, Mordasini L, Engeler DS. Prostatic Artery Embolisation Versus Transurethral Resection of the Prostate for Benign Prostatic Hyperplasia: 2-yr Outcomes of a Randomised, Open-label, Single-centre Trial. Eur Urol. 2021 Jul;80(1):34-42. doi: 10.1016/j.eururo.2021.02.008. Epub 2021 Feb 19. PMID 33612376
- [Derived] Mullhaupt G, Hechelhammer L, Graf N, Mordasini L, Schmid HP, Engeler DS, Abt D. Prostatic Artery Embolisation Versus Transurethral Resection of the Prostate for Benign Prostatic Obstruction: 5-year Outcomes of a Randomised, Open-label, Noninferiority Trial. Eur Urol Focus. 2024 Sep;10(5):788-795. doi: 10.1016/j.euf.2024.03.001. Epub 2024 Mar 25. PMID 38531756